CLINICAL TRIAL: NCT01803737
Title: Feasibility of a Campaign Intervention Compared to a Standard Behavioral Weight Loss Intervention in Overweight and Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, David Garcia, Doctoral Student, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO12110211
Record Dates: First submitted 2013-02-28; First posted 2013-03-04 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-01

CONDITIONS: Weight Loss
Keywords: Weight Loss; Physical Activity; Dietary Intake; Weight Loss Self-Efficacy; Motivation
MeSH Terms: conditions — Weight Loss; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Behavioral Weight Loss Intervention (SBWL) (Active Comparator): Included changing eating behaviors, increasing physical activity, and attending regular group weight loss meetings.
  Interventions: Behavioral: Standard Behavioral Weight Loss Intervention (SBWL)
- Campaign Intervention (CI) (Experimental): Included changing eating behaviors and increasing physical activity, however participants will not attend regular meetings. Instead they will attend two weekly meetings at weeks 0 and 12. During the weeks they are not scheduled to attend in-person weekly meetings (weeks 1-11), they will receive education materials via e-mail. They will also have the opportunity to earn points towards prizes by reporting diet and physical activity behaviors, and body weight via e-mail.
  Interventions: Behavioral: Campaign Intervention (CI)

INTERVENTIONS:
Behavioral: Standard Behavioral Weight Loss Intervention (SBWL) — Included changing eating behaviors, increasing physical activity, and attending regular group weight loss meetings.
  Arms: Standard Behavioral Weight Loss Intervention (SBWL)
Behavioral: Campaign Intervention (CI) — Included changing eating behaviors and increasing physical activity, however participants will not attend regular meetings. Instead they will attend two weekly meetings at weeks 0 and 12. During the weeks they are not scheduled to attend in-person weekly meetings (weeks 1-11), they will receive education materials via e-mail. They will also have the opportunity to earn points towards prizes by reporting diet and physical activity behaviors, and body weight via e-mail.
  Arms: Campaign Intervention (CI)

SUMMARY:
The purpose of this study is to examine the feasibility of a campaign intervention for weight management compared to a standard behavioral weight loss intervention in overweight and obese adults.

DETAILED DESCRIPTION:
The feasibility of solely using a campaign intervention (CI) to promote healthy eating and physical activity behaviors for weight loss and weight maintenance has not been examined in a systematic manner. Thus, the primary aim of this study will be to examine whether a stand-alone CI results in similar weight loss compared to a standard behavioral weight loss intervention (SBWL). It is hypothesized that the CI will achieve a similar weight loss when compared to the SBWL. Additional aims include the examination of the CI on changes in moderate to vigorous intensity physical activity, dietary intake, self-monitoring of dietary intake and physical activity, weight loss self-efficacy, and motivation compared to a SBWL. This study will recruit forty-eight sedentary, overweight and obese adult men and women, to participate in a behavioral weight loss intervention at the University of Pittsburgh Physical Activity and Weight Management Research Center (PAWMRC). To be considered eligible for this study, participants must be 18-55 years of age, with a Body Mass Index (BMI) ranging from ≥25.0 kg/m² to 45.0 kg/m². Assessments will be conducted at week 0 and 12 of the intervention. Each assessment will take approximately 30 minutes to complete and include height, body weight, and assessment of physical activity, dietary intake, weight loss self-efficacy, and motivation. Upon successful completion of baseline assessments, eligible subjects will be randomly assigned to one of two groups using a stratified randomized block design: 1) standard behavioral weight loss intervention (SBWL) or 2) campaign intervention (CI). The CI will target specific diet and physical activity behaviors to improve weight loss efforts within a thematic framework based on the professional auto racing point system concept. CI session content and targeted behavior goals will tie into this overall theme and throughout the campaign participants will have the opportunity to earn incentives to reinforce positive behavior changes. This study is a necessary first step to examine the feasibility of a stand-alone campaign as an alternative strategy for weight management when compared to a standard behavioral weight loss intervention. Furthermore, this study will provide variance estimates on the effectiveness of a campaign intervention compared to a standard behavioral weight loss program that can be used to determine appropriate sample sizes for a future full-scale clinical study of this alternative strategy.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years of age
* Body mass index (BMI) ranging from ≥25.0 kg/m² to 45.0 kg/m²
* Ability to provide informed consent

Exclusion Criteria:

* Regular exercise participation of at least 20 minutes per day on at least 3 days per week during the previous six months.
* Participation in a previous physical activity or weight management research project in the previous 6 months.
* Weight loss of ≥5% of current body weight in the previous 6 months.
* For women, those currently pregnant, pregnant during the previous 6 months, or plan on becoming pregnant in the next 6 months.
* History of myocardial infarction, coronary bypass surgery, angioplasty, or other heart-related surgeries.
* History of orthopedic or physical complications that would prevent participation in exercise.
* Currently taking any prescription medication that may affect metabolism and/or body weight (e.g., synthroid).
* Currently being treated for any condition that could affect body weight, such as coronary heart disease, diabetes mellitus, uncontrolled hypertension, cancer, depression, and anxiety.
* Currently being treated for any psychological issues or problems, taking any psychotropic medications, or receiving treatment with psychotropic medications within the previous 6 months.
* Resting systolic blood pressure ≥150mmHg or diastolic blood pressure ≥100mmHg. Subjects with controlled hypertension will be allowed to participate if they obtain a medical doctor's written consent to ensure that it is safe to participate in a weight loss intervention.
* Currently do not have access to a computer and the Internet.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David O Garcia, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Physical Activity and Weight Management Research Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Flegal KM, Carroll MD, Kit BK, Ogden CL. Prevalence of obesity and trends in the distribution of body mass index among US adults, 1999-2010. JAMA. 2012 Feb 1;307(5):491-7. doi: 10.1001/jama.2012.39. Epub 2012 Jan 17. PMID 22253363
- [Background] Cohen SS, Signorello LB, Cope EL, McLaughlin JK, Hargreaves MK, Zheng W, Blot WJ. Obesity and all-cause mortality among black adults and white adults. Am J Epidemiol. 2012 Sep 1;176(5):431-42. doi: 10.1093/aje/kws032. Epub 2012 Jul 20. PMID 22822174
- [Background] Pi-Sunyer FX. The obesity epidemic: pathophysiology and consequences of obesity. Obes Res. 2002 Dec;10 Suppl 2:97S-104S. doi: 10.1038/oby.2002.202. PMID 12490658
- [Background] Finkelstein EA, Trogdon JG, Cohen JW, Dietz W. Annual medical spending attributable to obesity: payer-and service-specific estimates. Health Aff (Millwood). 2009 Sep-Oct;28(5):w822-31. doi: 10.1377/hlthaff.28.5.w822. Epub 2009 Jul 27. PMID 19635784
- [Background] Clinical Guidelines on the Identification, Evaluation, and Treatment of Overweight and Obesity in Adults--The Evidence Report. National Institutes of Health. Obes Res. 1998 Sep;6 Suppl 2:51S-209S. No abstract available. PMID 9813653
- [Background] Berkel LA, Poston WS, Reeves RS, Foreyt JP. Behavioral interventions for obesity. J Am Diet Assoc. 2005 May;105(5 Suppl 1):S35-43. doi: 10.1016/j.jada.2005.02.031. PMID 15867894
- [Background] Look AHEAD Research Group; Wadden TA, West DS, Delahanty L, Jakicic J, Rejeski J, Williamson D, Berkowitz RI, Kelley DE, Tomchee C, Hill JO, Kumanyika S. The Look AHEAD study: a description of the lifestyle intervention and the evidence supporting it. Obesity (Silver Spring). 2006 May;14(5):737-52. doi: 10.1038/oby.2006.84. PMID 16855180
- [Background] Unick JL, Jakicic JM, Marcus BH. Contribution of behavior intervention components to 24-month weight loss. Med Sci Sports Exerc. 2010 Apr;42(4):745-53. doi: 10.1249/MSS.0b013e3181bd1a57. PMID 19952841
- [Background] Donnelly JE, Blair SN, Jakicic JM, Manore MM, Rankin JW, Smith BK; American College of Sports Medicine. American College of Sports Medicine Position Stand. Appropriate physical activity intervention strategies for weight loss and prevention of weight regain for adults. Med Sci Sports Exerc. 2009 Feb;41(2):459-71. doi: 10.1249/MSS.0b013e3181949333. PMID 19127177
- [Background] Jakicic JM, Tate DF, Lang W, Davis KK, Polzien K, Rickman AD, Erickson K, Neiberg RH, Finkelstein EA. Effect of a stepped-care intervention approach on weight loss in adults: a randomized clinical trial. JAMA. 2012 Jun 27;307(24):2617-26. doi: 10.1001/jama.2012.6866. PMID 22735431
- [Background] Diabetes Prevention Program (DPP) Research Group. The Diabetes Prevention Program (DPP): description of lifestyle intervention. Diabetes Care. 2002 Dec;25(12):2165-71. doi: 10.2337/diacare.25.12.2165. PMID 12453955
- [Background] Hamman RF, Wing RR, Edelstein SL, Lachin JM, Bray GA, Delahanty L, Hoskin M, Kriska AM, Mayer-Davis EJ, Pi-Sunyer X, Regensteiner J, Venditti B, Wylie-Rosett J. Effect of weight loss with lifestyle intervention on risk of diabetes. Diabetes Care. 2006 Sep;29(9):2102-7. doi: 10.2337/dc06-0560. PMID 16936160
- [Background] Look AHEAD Research Group; Pi-Sunyer X, Blackburn G, Brancati FL, Bray GA, Bright R, Clark JM, Curtis JM, Espeland MA, Foreyt JP, Graves K, Haffner SM, Harrison B, Hill JO, Horton ES, Jakicic J, Jeffery RW, Johnson KC, Kahn S, Kelley DE, Kitabchi AE, Knowler WC, Lewis CE, Maschak-Carey BJ, Montgomery B, Nathan DM, Patricio J, Peters A, Redmon JB, Reeves RS, Ryan DH, Safford M, Van Dorsten B, Wadden TA, Wagenknecht L, Wesche-Thobaben J, Wing RR, Yanovski SZ. Reduction in weight and cardiovascular disease risk factors in individuals with type 2 diabetes: one-year results of the look AHEAD trial. Diabetes Care. 2007 Jun;30(6):1374-83. doi: 10.2337/dc07-0048. Epub 2007 Mar 15. PMID 17363746
- [Background] Obesity: preventing and managing the global epidemic. Report of a WHO consultation. World Health Organ Tech Rep Ser. 2000;894:i-xii, 1-253. PMID 11234459
- [Background] Wadden TA, Crerand CE, Brock J. Behavioral treatment of obesity. Psychiatr Clin North Am. 2005 Mar;28(1):151-70, ix. doi: 10.1016/j.psc.2004.09.008. No abstract available. PMID 15733617
- [Background] Levy RL, Finch EA, Crowell MD, Talley NJ, Jeffery RW. Behavioral intervention for the treatment of obesity: strategies and effectiveness data. Am J Gastroenterol. 2007 Oct;102(10):2314-21. doi: 10.1111/j.1572-0241.2007.01342.x. Epub 2007 Jun 11. PMID 17561967
- [Background] Pearson ES. Goal setting as a health behavior change strategy in overweight and obese adults: a systematic literature review examining intervention components. Patient Educ Couns. 2012 Apr;87(1):32-42. doi: 10.1016/j.pec.2011.07.018. Epub 2011 Aug 17. PMID 21852063
- [Background] Volpp KG, John LK, Troxel AB, Norton L, Fassbender J, Loewenstein G. Financial incentive-based approaches for weight loss: a randomized trial. JAMA. 2008 Dec 10;300(22):2631-7. doi: 10.1001/jama.2008.804. PMID 19066383
- [Background] Foster GD, Makris AP, Bailer BA. Behavioral treatment of obesity. Am J Clin Nutr. 2005 Jul;82(1 Suppl):230S-235S. doi: 10.1093/ajcn/82.1.230S. PMID 16002827
- [Background] Locke EA, Latham GP. Building a practically useful theory of goal setting and task motivation. A 35-year odyssey. Am Psychol. 2002 Sep;57(9):705-17. doi: 10.1037//0003-066x.57.9.705. PMID 12237980
- [Background] Nothwehr F, Yang J. Goal setting frequency and the use of behavioral strategies related to diet and physical activity. Health Educ Res. 2007 Aug;22(4):532-8. doi: 10.1093/her/cyl117. Epub 2006 Oct 10. PMID 17032703
- [Background] Dubbert PM, Wilson GT. Goal-setting and spouse involvement in the treatment of obesity. Behav Res Ther. 1984;22(3):227-42. doi: 10.1016/0005-7967(84)90003-2. No abstract available. PMID 6466273
- [Background] Bandura A. Social cognitive theory: an agentic perspective. Annu Rev Psychol. 2001;52:1-26. doi: 10.1146/annurev.psych.52.1.1. PMID 11148297
- [Background] Burke LE, Wang J, Sevick MA. Self-monitoring in weight loss: a systematic review of the literature. J Am Diet Assoc. 2011 Jan;111(1):92-102. doi: 10.1016/j.jada.2010.10.008. PMID 21185970
- [Background] Butryn ML, Phelan S, Hill JO, Wing RR. Consistent self-monitoring of weight: a key component of successful weight loss maintenance. Obesity (Silver Spring). 2007 Dec;15(12):3091-6. doi: 10.1038/oby.2007.368. PMID 18198319
- [Background] Helsel DL, Jakicic JM, Otto AD. Comparison of techniques for self-monitoring eating and exercise behaviors on weight loss in a correspondence-based intervention. J Am Diet Assoc. 2007 Oct;107(10):1807-10. doi: 10.1016/j.jada.2007.07.014. PMID 17904942
- [Background] Wadden TA, Berkowitz RI, Womble LG, Sarwer DB, Phelan S, Cato RK, Hesson LA, Osei SY, Kaplan R, Stunkard AJ. Randomized trial of lifestyle modification and pharmacotherapy for obesity. N Engl J Med. 2005 Nov 17;353(20):2111-20. doi: 10.1056/NEJMoa050156. PMID 16291981
- [Background] Boutelle KN, Kirschenbaum DS, Baker RC, Mitchell ME. How can obese weight controllers minimize weight gain during the high risk holiday season? By self-monitoring very consistently. Health Psychol. 1999 Jul;18(4):364-8. doi: 10.1037//0278-6133.18.4.364. PMID 10431937
- [Background] Burke LE, Conroy MB, Sereika SM, Elci OU, Styn MA, Acharya SD, Sevick MA, Ewing LJ, Glanz K. The effect of electronic self-monitoring on weight loss and dietary intake: a randomized behavioral weight loss trial. Obesity (Silver Spring). 2011 Feb;19(2):338-44. doi: 10.1038/oby.2010.208. Epub 2010 Sep 16. PMID 20847736
- [Background] Tate DF, Wing RR, Winett RA. Using Internet technology to deliver a behavioral weight loss program. JAMA. 2001 Mar 7;285(9):1172-7. doi: 10.1001/jama.285.9.1172. PMID 11231746
- [Background] Wing RR, Crane MM, Thomas JG, Kumar R, Weinberg B. Improving weight loss outcomes of community interventions by incorporating behavioral strategies. Am J Public Health. 2010 Dec;100(12):2513-9. doi: 10.2105/AJPH.2009.183616. Epub 2010 Oct 21. PMID 20966375
- [Background] Wing RR. Behavioral treatment of severe obesity. Am J Clin Nutr. 1992 Feb;55(2 Suppl):545S-551S. doi: 10.1093/ajcn/55.2.545s. PMID 1733124
- [Background] Butsch WS, Ard JD, Allison DB, Patki A, Henson CS, Rueger MM, Hubbert KA, Glandon GL, Heimburger DC. Effects of a reimbursement incentive on enrollment in a weight control program. Obesity (Silver Spring). 2007 Nov;15(11):2733-8. doi: 10.1038/oby.2007.325. PMID 18070764
- [Background] Jeffery RW, Wing RR, Thorson C, Burton LR, Raether C, Harvey J, Mullen M. Strengthening behavioral interventions for weight loss: a randomized trial of food provision and monetary incentives. J Consult Clin Psychol. 1993 Dec;61(6):1038-45. doi: 10.1037//0022-006x.61.6.1038. PMID 8113481
- [Background] Jeffery RW, Wing RR. Long-term effects of interventions for weight loss using food provision and monetary incentives. J Consult Clin Psychol. 1995 Oct;63(5):793-6. doi: 10.1037//0022-006x.63.5.793. PMID 7593872
- [Background] Jeffery RW, Gerber WM, Rosenthal BS, Lindquist RA. Monetary contracts in weight control: effectiveness of group and individual contracts of varying size. J Consult Clin Psychol. 1983 Apr;51(2):242-8. doi: 10.1037//0022-006x.51.2.242. No abstract available. PMID 6841768
- [Background] Jeffery RW, Wing RR, Thorson C, Burton LR. Use of personal trainers and financial incentives to increase exercise in a behavioral weight-loss program. J Consult Clin Psychol. 1998 Oct;66(5):777-83. doi: 10.1037//0022-006x.66.5.777. PMID 9803696
- [Background] Jeffery RW, Thompson PD, Wing RR. Effects on weight reduction of strong monetary contracts for calorie restriction or weight loss. Behav Res Ther. 1978;16(5):363-9. doi: 10.1016/0005-7967(78)90005-0. No abstract available. PMID 743075
- [Background] Ryan RM, Deci EL. Self-determination theory and the facilitation of intrinsic motivation, social development, and well-being. Am Psychol. 2000 Jan;55(1):68-78. doi: 10.1037//0003-066x.55.1.68. PMID 11392867
- [Background] Deci EL, Ryan RM. The support of autonomy and the control of behavior. J Pers Soc Psychol. 1987 Dec;53(6):1024-37. doi: 10.1037//0022-3514.53.6.1024. PMID 3320334
- [Background] Carton JS. The differential effects of tangible rewards and praise on intrinsic motivation: A comparison of cognitive evaluation theory and operant theory. Behav Anal. 1996 Fall;19(2):237-55. doi: 10.1007/BF03393167. PMID 22478261
- [Background] Crane MM, Tate DF, Finkelstein EA, Linnan LA. Motivation for participating in a weight loss program and financial incentives: an analysis from a randomized trial. J Obes. 2012;2012:290589. doi: 10.1155/2012/290589. Epub 2012 Apr 17. PMID 22577524
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of obesity and trends in body mass index among US children and adolescents, 1999-2010. JAMA. 2012 Feb 1;307(5):483-90. doi: 10.1001/jama.2012.40. Epub 2012 Jan 17. PMID 22253364
- [Background] Wadden TA, Butryn ML, Wilson C. Lifestyle modification for the management of obesity. Gastroenterology. 2007 May;132(6):2226-38. doi: 10.1053/j.gastro.2007.03.051. PMID 17498514
- [Background] Curioni CC, Lourenco PM. Long-term weight loss after diet and exercise: a systematic review. Int J Obes (Lond). 2005 Oct;29(10):1168-74. doi: 10.1038/sj.ijo.0803015. PMID 15925949
- [Background] Flegal KM, Carroll MD, Kuczmarski RJ, Johnson CL. Overweight and obesity in the United States: prevalence and trends, 1960-1994. Int J Obes Relat Metab Disord. 1998 Jan;22(1):39-47. doi: 10.1038/sj.ijo.0800541. PMID 9481598
- [Background] Flegal KM, Carroll MD, Ogden CL, Johnson CL. Prevalence and trends in obesity among US adults, 1999-2000. JAMA. 2002 Oct 9;288(14):1723-7. doi: 10.1001/jama.288.14.1723. PMID 12365955
- [Background] Klein S, Burke LE, Bray GA, Blair S, Allison DB, Pi-Sunyer X, Hong Y, Eckel RH; American Heart Association Council on Nutrition, Physical Activity, and Metabolism. Clinical implications of obesity with specific focus on cardiovascular disease: a statement for professionals from the American Heart Association Council on Nutrition, Physical Activity, and Metabolism: endorsed by the American College of Cardiology Foundation. Circulation. 2004 Nov 2;110(18):2952-67. doi: 10.1161/01.CIR.0000145546.97738.1E. Epub 2004 Oct 27. PMID 15509809
- [Background] Field AE, Coakley EH, Must A, Spadano JL, Laird N, Dietz WH, Rimm E, Colditz GA. Impact of overweight on the risk of developing common chronic diseases during a 10-year period. Arch Intern Med. 2001 Jul 9;161(13):1581-6. doi: 10.1001/archinte.161.13.1581. PMID 11434789
- [Background] Flegal KM, Graubard BI, Williamson DF, Gail MH. Excess deaths associated with underweight, overweight, and obesity. JAMA. 2005 Apr 20;293(15):1861-7. doi: 10.1001/jama.293.15.1861. PMID 15840860
- [Background] Finkelstein EA, Fiebelkorn IC, Wang G. National medical spending attributable to overweight and obesity: how much, and who's paying? Health Aff (Millwood). 2003 Jan-Jun;Suppl Web Exclusives:W3-219-26. doi: 10.1377/hlthaff.w3.219. PMID 14527256
- [Background] Ostbye T, Dement JM, Krause KM. Obesity and workers' compensation: results from the Duke Health and Safety Surveillance System. Arch Intern Med. 2007 Apr 23;167(8):766-73. doi: 10.1001/archinte.167.8.766. PMID 17452538
- [Background] Tucker LA, Friedman GM. Obesity and absenteeism: an epidemiologic study of 10,825 employed adults. Am J Health Promot. 1998 Jan-Feb;12(3):202-7. doi: 10.4278/0890-1171-12.3.202. PMID 10176095
- [Background] Finkelstein EA, DiBonaventura Md, Burgess SM, Hale BC. The costs of obesity in the workplace. J Occup Environ Med. 2010 Oct;52(10):971-6. doi: 10.1097/JOM.0b013e3181f274d2. PMID 20881629
- [Background] Mitchell NS, Catenacci VA, Wyatt HR, Hill JO. Obesity: overview of an epidemic. Psychiatr Clin North Am. 2011 Dec;34(4):717-32. doi: 10.1016/j.psc.2011.08.005. PMID 22098799
- [Background] Peters JC, Wyatt HR, Donahoo WT, Hill JO. From instinct to intellect: the challenge of maintaining healthy weight in the modern world. Obes Rev. 2002 May;3(2):69-74. doi: 10.1046/j.1467-789x.2002.00059.x. PMID 12120422
- [Background] Hill JO, Wyatt HR, Melanson EL. Genetic and environmental contributions to obesity. Med Clin North Am. 2000 Mar;84(2):333-46. doi: 10.1016/s0025-7125(05)70224-8. PMID 10793645
- [Background] Hill JO, Wyatt HR, Peters JC. Energy balance and obesity. Circulation. 2012 Jul 3;126(1):126-32. doi: 10.1161/CIRCULATIONAHA.111.087213. PMID 22753534
- [Background] Pender JR, Pories WJ. Epidemiology of obesity in the United States. Gastroenterol Clin North Am. 2005 Mar;34(1):1-7. doi: 10.1016/j.gtc.2004.12.010. PMID 15823434
- [Background] Bouchard C. Defining the genetic architecture of the predisposition to obesity: a challenging but not insurmountable task. Am J Clin Nutr. 2010 Jan;91(1):5-6. doi: 10.3945/ajcn.2009.28933. Epub 2009 Nov 25. No abstract available. PMID 19939981
- [Background] Hill JO, Wyatt HR, Reed GW, Peters JC. Obesity and the environment: where do we go from here? Science. 2003 Feb 7;299(5608):853-5. doi: 10.1126/science.1079857. PMID 12574618
- [Background] Butryn ML, Webb V, Wadden TA. Behavioral treatment of obesity. Psychiatr Clin North Am. 2011 Dec;34(4):841-59. doi: 10.1016/j.psc.2011.08.006. PMID 22098808
- [Background] Poston WS 2nd, Foreyt JP. Successful management of the obese patient. Am Fam Physician. 2000 Jun 15;61(12):3615-22. PMID 10892633
- [Background] United States Department of Health and Human Services. Dietary Guidelines for Americans, 2010. http://www.cnpp.usda.gov/DGAs2010-PolicyDocument.htm. Accessed August 14, 2012.
- [Background] Tsai AG, Wadden TA. The evolution of very-low-calorie diets: an update and meta-analysis. Obesity (Silver Spring). 2006 Aug;14(8):1283-93. doi: 10.1038/oby.2006.146. PMID 16988070
- [Background] Ditschuneit HH, Flechtner-Mors M, Johnson TD, Adler G. Metabolic and weight-loss effects of a long-term dietary intervention in obese patients. Am J Clin Nutr. 1999 Feb;69(2):198-204. doi: 10.1093/ajcn/69.2.198. PMID 9989680
- [Background] Flechtner-Mors M, Ditschuneit HH, Johnson TD, Suchard MA, Adler G. Metabolic and weight loss effects of long-term dietary intervention in obese patients: four-year results. Obes Res. 2000 Aug;8(5):399-402. doi: 10.1038/oby.2000.48. PMID 10968732
- [Background] Heymsfield SB, van Mierlo CA, van der Knaap HC, Heo M, Frier HI. Weight management using a meal replacement strategy: meta and pooling analysis from six studies. Int J Obes Relat Metab Disord. 2003 May;27(5):537-49. doi: 10.1038/sj.ijo.0802258. PMID 12704397
- [Background] Wing RR, Jeffery RW, Burton LR, Thorson C, Nissinoff KS, Baxter JE. Food provision vs structured meal plans in the behavioral treatment of obesity. Int J Obes Relat Metab Disord. 1996 Jan;20(1):56-62. PMID 8788323
- [Background] Caspersen CJ, Powell KE, Christenson GM. Physical activity, exercise, and physical fitness: definitions and distinctions for health-related research. Public Health Rep. 1985 Mar-Apr;100(2):126-31. PMID 3920711
- [Background] Pate RR, Pratt M, Blair SN, Haskell WL, Macera CA, Bouchard C, Buchner D, Ettinger W, Heath GW, King AC, et al. Physical activity and public health. A recommendation from the Centers for Disease Control and Prevention and the American College of Sports Medicine. JAMA. 1995 Feb 1;273(5):402-7. doi: 10.1001/jama.273.5.402. PMID 7823386
- [Background] Donnelly JE, Smith B, Jacobsen DJ, Kirk E, Dubose K, Hyder M, Bailey B, Washburn R. The role of exercise for weight loss and maintenance. Best Pract Res Clin Gastroenterol. 2004 Dec;18(6):1009-29. doi: 10.1016/j.bpg.2004.06.022. PMID 15561636
- [Background] Jakicic JM, Clark K, Coleman E, Donnelly JE, Foreyt J, Melanson E, Volek J, Volpe SL; American College of Sports Medicine. American College of Sports Medicine position stand. Appropriate intervention strategies for weight loss and prevention of weight regain for adults. Med Sci Sports Exerc. 2001 Dec;33(12):2145-56. doi: 10.1097/00005768-200112000-00026. PMID 11740312
- [Background] Weyer C, Linkeschowa R, Heise T, Giesen HT, Spraul M. Implications of the traditional and the new ACSM physical activity recommendations on weight reduction in dietary treated obese subjects. Int J Obes Relat Metab Disord. 1998 Nov;22(11):1071-8. doi: 10.1038/sj.ijo.0800728. PMID 9822944
- [Background] Hill JO, Wyatt HR. Role of physical activity in preventing and treating obesity. J Appl Physiol (1985). 2005 Aug;99(2):765-70. doi: 10.1152/japplphysiol.00137.2005. PMID 16020440
- [Background] Catenacci VA, Wyatt HR. The role of physical activity in producing and maintaining weight loss. Nat Clin Pract Endocrinol Metab. 2007 Jul;3(7):518-29. doi: 10.1038/ncpendmet0554. PMID 17581621
- [Background] Jakicic JM, Davis KK. Obesity and physical activity. Psychiatr Clin North Am. 2011 Dec;34(4):829-40. doi: 10.1016/j.psc.2011.08.009. Epub 2011 Oct 15. PMID 22098807
- [Background] Miller WC, Koceja DM, Hamilton EJ. A meta-analysis of the past 25 years of weight loss research using diet, exercise or diet plus exercise intervention. Int J Obes Relat Metab Disord. 1997 Oct;21(10):941-7. doi: 10.1038/sj.ijo.0800499. PMID 9347414
- [Background] Wing RR. Physical activity in the treatment of the adulthood overweight and obesity: current evidence and research issues. Med Sci Sports Exerc. 1999 Nov;31(11 Suppl):S547-52. doi: 10.1097/00005768-199911001-00010. PMID 10593526
- [Background] Slentz CA, Duscha BD, Johnson JL, Ketchum K, Aiken LB, Samsa GP, Houmard JA, Bales CW, Kraus WE. Effects of the amount of exercise on body weight, body composition, and measures of central obesity: STRRIDE--a randomized controlled study. Arch Intern Med. 2004 Jan 12;164(1):31-9. doi: 10.1001/archinte.164.1.31. PMID 14718319
- [Background] Jeffery RW, Wing RR, Sherwood NE, Tate DF. Physical activity and weight loss: does prescribing higher physical activity goals improve outcome? Am J Clin Nutr. 2003 Oct;78(4):684-9. doi: 10.1093/ajcn/78.4.684. PMID 14522725
- [Background] Jakicic JM, Marcus BH, Lang W, Janney C. Effect of exercise on 24-month weight loss maintenance in overweight women. Arch Intern Med. 2008 Jul 28;168(14):1550-9; discussion 1559-60. doi: 10.1001/archinte.168.14.1550. PMID 18663167
- [Background] Shilts MK, Horowitz M, Townsend MS. Goal setting as a strategy for dietary and physical activity behavior change: a review of the literature. Am J Health Promot. 2004 Nov-Dec;19(2):81-93. doi: 10.4278/0890-1171-19.2.81. PMID 15559708
- [Background] Schneider PL, Bassett DR Jr, Thompson DL, Pronk NP, Bielak KM. Effects of a 10,000 steps per day goal in overweight adults. Am J Health Promot. 2006 Nov-Dec;21(2):85-9. doi: 10.4278/0890-1171-21.2.85. PMID 17152246
- [Background] Schnoll R, Zimmerman BJ. Self-regulation training enhances dietary self-efficacy and dietary fiber consumption. J Am Diet Assoc. 2001 Sep;101(9):1006-11. doi: 10.1016/S0002-8223(01)00249-8. PMID 11573751
- [Background] Bodenheimer T, Handley MA. Goal-setting for behavior change in primary care: an exploration and status report. Patient Educ Couns. 2009 Aug;76(2):174-80. doi: 10.1016/j.pec.2009.06.001. Epub 2009 Jun 27. PMID 19560895
- [Background] Boutelle KN, Kirschenbaum DS. Further support for consistent self-monitoring as a vital component of successful weight control. Obes Res. 1998 May;6(3):219-24. doi: 10.1002/j.1550-8528.1998.tb00340.x. PMID 9618126
- [Background] Linde JA, Jeffery RW, French SA, Pronk NP, Boyle RG. Self-weighing in weight gain prevention and weight loss trials. Ann Behav Med. 2005 Dec;30(3):210-6. doi: 10.1207/s15324796abm3003_5. PMID 16336072
- [Background] Strecher VJ, Seijts GH, Kok GJ, Latham GP, Glasgow R, DeVellis B, Meertens RM, Bulger DW. Goal setting as a strategy for health behavior change. Health Educ Q. 1995 May;22(2):190-200. doi: 10.1177/109019819502200207. PMID 7622387
- [Background] Tate DF, Jackvony EH, Wing RR. A randomized trial comparing human e-mail counseling, computer-automated tailored counseling, and no counseling in an Internet weight loss program. Arch Intern Med. 2006 Aug 14-28;166(15):1620-5. doi: 10.1001/archinte.166.15.1620. PMID 16908795
- [Background] United States Census Bureau. Computer and Internet Use. 2010 http://www.census.gov/hhes/computer/1. Accessed November 12, 2012.
- [Background] Kodama S, Saito K, Tanaka S, Horikawa C, Fujiwara K, Hirasawa R, Yachi Y, Iida KT, Shimano H, Ohashi Y, Yamada N, Sone H. Effect of Web-based lifestyle modification on weight control: a meta-analysis. Int J Obes (Lond). 2012 May;36(5):675-85. doi: 10.1038/ijo.2011.121. Epub 2011 Jun 21. PMID 21694698
- [Background] Jeffery RW, Drewnowski A, Epstein LH, Stunkard AJ, Wilson GT, Wing RR, Hill DR. Long-term maintenance of weight loss: current status. Health Psychol. 2000 Jan;19(1S):5-16. doi: 10.1037/0278-6133.19.suppl1.5. PMID 10709944
- [Background] Finkelstein EA, Linnan LA, Tate DF, Birken BE. A pilot study testing the effect of different levels of financial incentives on weight loss among overweight employees. J Occup Environ Med. 2007 Sep;49(9):981-9. doi: 10.1097/JOM.0b013e31813c6dcb. PMID 17848854
- [Background] Petry NM, Barry D, Pescatello L, White WB. A low-cost reinforcement procedure improves short-term weight loss outcomes. Am J Med. 2011 Nov;124(11):1082-5. doi: 10.1016/j.amjmed.2011.04.016. Epub 2011 Aug 17. PMID 21851917
- [Background] Elfhag K, Rossner S. Who succeeds in maintaining weight loss? A conceptual review of factors associated with weight loss maintenance and weight regain. Obes Rev. 2005 Feb;6(1):67-85. doi: 10.1111/j.1467-789X.2005.00170.x. PMID 15655039
- [Background] Williams GC, Grow VM, Freedman ZR, Ryan RM, Deci EL. Motivational predictors of weight loss and weight-loss maintenance. J Pers Soc Psychol. 1996 Jan;70(1):115-26. doi: 10.1037//0022-3514.70.1.115. PMID 8558405
- [Background] Wing RR, Gillis B. The Diabetes Prevention Program's Lifestyle Change Program Appendix G: Toolbox. [DPP Lifestyle Change Program Manual of Operations]. 1996; 1-123. Available at: http://www.bsc.gwu.edu/dpp/lifestyle/apndxg.pdf.
- [Background] Otto AD, Jakicic JM, Gallagher KI, Thomas EL, Mohr CR. Effect of an Incentive-Based Motivational Campaign on Weight Loss and Physical Activity in Overweight Women. Medicine & Science in Sports & Exercise. May 2004;36(5):S299-S300.
- [Background] Otto AD, Jakicic JM. Examination of usefulness of time-based strategies on weight loss and physical activity in overweight adults [Abstract]. Obesity (Silver Spring). 2007;15(9:Supplement).
- [Background] Canadian Society for Exercise Physiology. PAR-Q and You. 2002. http://www.csep.ca/cmfiles/publications/parq/par-q.pdf. Accessed August 14, 2012.
- [Background] D'Zurilla TJ, Goldfried MR. Problem solving and behavior modification. J Abnorm Psychol. 1971 Aug;78(1):107-26. doi: 10.1037/h0031360. No abstract available. PMID 4938262
- [Background] Borushek A. 2012 CalorieKing Calorie, Fat and Carbohydrate Counter: Costa Mesa, CA: Family Health Publications; 2012.
- [Background] Goss F, Robertson R, DaSilva S, Suminski R, Kang J, Metz K. Ratings of perceived exertion and energy expenditure during light to moderate activity. Percept Mot Skills. 2003 Jun;96(3 Pt 1):739-47. doi: 10.2466/pms.2003.96.3.739. PMID 12831247
- [Background] Bellg AJ, Borrelli B, Resnick B, Hecht J, Minicucci DS, Ory M, Ogedegbe G, Orwig D, Ernst D, Czajkowski S; Treatment Fidelity Workgroup of the NIH Behavior Change Consortium. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. Health Psychol. 2004 Sep;23(5):443-51. doi: 10.1037/0278-6133.23.5.443. PMID 15367063
- [Background] Block G, Hartman AM, Dresser CM, Carroll MD, Gannon J, Gardner L. A data-based approach to diet questionnaire design and testing. Am J Epidemiol. 1986 Sep;124(3):453-69. doi: 10.1093/oxfordjournals.aje.a114416. PMID 3740045
- [Background] Block G, Woods M, Potosky A, Clifford C. Validation of a self-administered diet history questionnaire using multiple diet records. J Clin Epidemiol. 1990;43(12):1327-35. doi: 10.1016/0895-4356(90)90099-b. PMID 2254769
- [Background] O'Neil PM, Rieder S. Utility and validity of the eating behavior inventory in clinical obesity research: a review of the literature. Obes Rev. 2005 Aug;6(3):209-16. doi: 10.1111/j.1467-789X.2005.00192.x. PMID 16045636
- [Background] Paffenbarger RS Jr, Hyde RT, Wing AL, Hsieh CC. Physical activity, all-cause mortality, and longevity of college alumni. N Engl J Med. 1986 Mar 6;314(10):605-13. doi: 10.1056/NEJM198603063141003. PMID 3945246
- [Background] Pereira MA, FitzerGerald SJ, Gregg EW, Joswiak ML, Ryan WJ, Suminski RR, Utter AC, Zmuda JM. A collection of Physical Activity Questionnaires for health-related research. Med Sci Sports Exerc. 1997 Jun;29(6 Suppl):S1-205. No abstract available. PMID 9243481
- [Background] Clark MM, Abrams DB, Niaura RS, Eaton CA, Rossi JS. Self-efficacy in weight management. J Consult Clin Psychol. 1991 Oct;59(5):739-44. doi: 10.1037//0022-006x.59.5.739. PMID 1955608
- [Background] Fontaine KR, Cheskin LJ. Self-efficacy, attendance, and weight loss in obesity treatment. Addict Behav. 1997 Jul-Aug;22(4):567-70. doi: 10.1016/s0306-4603(96)00068-8. PMID 9290865
- [Background] VanWormer JJ, Martinez AM, Cosentino D, Pronk NP. Satisfaction with a weight loss program: what matters? Am J Health Promot. 2010 Mar-Apr;24(4):238-45. doi: 10.4278/ajhp.080613-QUAN-92. PMID 20232605
- [Background] Baldwin AS, Rothman AJ, Jeffery RW. Satisfaction with weight loss: examining the longitudinal covariation between people's weight-loss-related outcomes and experiences and their satisfaction. Ann Behav Med. 2009 Dec;38(3):213-24. doi: 10.1007/s12160-009-9148-x. PMID 20082163

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited twenty six (N=26) sedentary, overweight and obese adult men and women to participate in a behavioral weight loss intervention at the University of Pittsburgh Physical Activity and Weight Management Research Center. Recruitment occurred between January 2013 and March 2013.
Groups:
- Standard Behavioral Weight Loss Intervention (SBWL): Includes changing eating behaviors, increasing physical activity, and attending regular group weight loss meetings.
- Campaign Intervention (CI): Includes changing eating behaviors and increasing physical activity, however participants will not attend regular meetings. Instead they will attend two weekly meetings at weeks 0 and 12. During the weeks they are not scheduled to attend in-person weekly meetings (weeks 1-11), they will receive education materials via e-mail. They will also have the opportunity to earn points towards prizes by reporting diet and physical activity behaviors, and body weight via e-mail.
Period: Overall Study
Arm/Group | Standard Behavioral Weight Loss Intervention (SBWL) | Campaign Intervention (CI)
Started | 13 | 13
Completed | 12 | 10
Not Completed | 1 | 3
Not completed — Lack of Time | 1 | 0
Not completed — Medical Reason | 0 | 1
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: Statistical analyses were performed using the Statistical Package for the Social Sciences (IBM-SPSS, version 21.0). Statistical significance was accepted at the p<0.05 level of confidence. Analyses were conducted using individuals who completed assessments at week 0 and 12, with intent-to-treat (ITT) analysis carrying the baseline data forward.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Behavioral Weight Loss Intervention (SBWL) | Campaign Intervention (CI) | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (9.1) | 43.8 (9.0) | 43.1 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: Body weight will be measured on a digital scale to assess change in body weight over the 12-week intervention period.
Time Frame: Week 0 and 12
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Standard Behavioral Weight Loss Intervention (SBWL) | Campaign Intervention (CI)
Number analyzed (Participants) | 13 | 13
kg | -5.6 (2.9) | -3.1 (3.4)

2. Secondary Outcome: Change in Physical Activity
Description: A questionnaire will be used to measure and quantify energy expenditure from physical activity.
Time Frame: Week 0 and 12
Measure: Mean (Standard Deviation); unit: kcals/wk
Arm/Group | Standard Behavioral Weight Loss Intervention (SBWL) | Campaign Intervention (CI)
Number analyzed (Participants) | 13 | 13
kcals/wk | 983.3 (567.6) | 776.3 (1194.8)

3. Secondary Outcome: Change in Dietary Intake: Kcals/Day
Description: A questionnaire will be used to assess self-reported food intake. This will be used to estimate calories, dietary fat, protein, and carbohydrates consumed.
Time Frame: Week 0 and 12
Measure: Mean (Standard Deviation); unit: kcals/day
Arm/Group | Standard Behavioral Weight Loss Intervention (SBWL) | Campaign Intervention (CI)
Number analyzed (Participants) | 13 | 13
kcals/day | 474.8 (509) | 242.5 (709.3)

4. Secondary Outcome: Change in Dietary Intake: % Fat
Description: as for outcome 3
Time Frame: Week 0 and 12
Measure: Mean (Standard Deviation); unit: percentage of fat intake
Arm/Group | Standard Behavioral Weight Loss Intervention (SBWL) | Campaign Intervention (CI)
Number analyzed (Participants) | 13 | 13
percentage of fat intake | -3.26 (5.58) | -0.00 (4.27)

5. Secondary Outcome: Change in Dietary Intake: % Protein
Description: as for outcome 3
Time Frame: Week 0 and 12
Measure: Mean (Standard Deviation); unit: percentage of protein intake
Arm/Group | Standard Behavioral Weight Loss Intervention (SBWL) | Campaign Intervention (CI)
Number analyzed (Participants) | 13 | 13
percentage of protein intake | 0.73 (2.38) | 0.44 (2.57)

6. Secondary Outcome: Change in Dietary Intake: % Carbohydrate
Description: as for outcome 3
Time Frame: Week 0 and 12
Measure: Mean (Standard Deviation); unit: percentage of carbohydrate intake
Arm/Group | Standard Behavioral Weight Loss Intervention (SBWL) | Campaign Intervention (CI)
Number analyzed (Participants) | 13 | 13
percentage of carbohydrate intake | 0.64 (6.15) | 0.90 (5.24)

7. Secondary Outcome: Completion of Self-monitoring of Dietary Intake and Physical Activity
Description: The frequency that participants engaged in the self-monitoring of dietary intake and physical activity was assessed at week 12. The diaries were completed weekly throughout the study.
Time Frame: Week 0 and 12
Measure: Mean (Standard Deviation); unit: percentage of diaries completed
Units Other Than Participants: Eating and Exercise Diary
Arm/Group | Standard Behavioral Weight Loss Intervention (SBWL) | Campaign Intervention (CI)
Number analyzed (Participants) | 13 | 13
Number analyzed (Eating and Exercise Diary) | 143 | 143
percentage of diaries completed | 91.6 (18) | 60.1 (38.5)

8. Secondary Outcome: Change in Weight Loss Self-efficacy
Description: Self-efficacy for weight loss was assessed at week 0 and 12 using a 20-item Weight Efficacy Lifestyle Questionnaire (WEL). The total score ranges from 0-180. Higher values represent greater beliefs toward the completion of weight management behaviors.
Time Frame: Week 0 and 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Behavioral Weight Loss Intervention (SBWL) | Campaign Intervention (CI)
Number analyzed (Participants) | 13 | 13
units on a scale | 28.3 (35.7) | 16.3 (35.8)

9. Secondary Outcome: Autonomous and Controlled Motivation
Description: At week 12, participants completed the 13-item TSRQ to assess motivation to continue to participate in the program if given the opportunity. The TSRQ represents participants' reasons for continuing participation in a weight loss program via participants' endorsement of statements of autonomous and controlled motivation. Responses were given using a 7-point Likert scale (1 = not at all true to 7 = very true). The responses on the autonomous items (5) and controlled items (8) were averaged.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Behavioral Weight Loss Intervention (SBWL) | Campaign Intervention (CI)
Number analyzed (Participants) | 12 | 10
units on a scale
  Autonomous Motivation | 6.3 (0.9) | 5.3 (1.5)
  Controlled Motivation | 2.9 (1.1) | 2.9 (1.0)

ADVERSE EVENTS:
Arm/Group | Standard Behavioral Weight Loss Intervention (SBWL) | Campaign Intervention (CI)
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes